CLINICAL TRIAL: NCT03224286
Title: Pressure Sensitive Mats for Patient Monitoring in the NICU
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: NSERC Collaborative Research and Development (Unknown)
Responsible Party: Principal Investigator, JoAnn Harrold, Division Chief, Neonatology, Children's Hospital of Eastern Ontario
Other Study IDs: REB#17/76X
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Apnea; Respiration Disorder
Keywords: Pressure sensitive mat
MeSH Terms: conditions — Apnea; Respiration Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Incubator + <1500 g: Infants currently in an incubator with a weight of less than 1500 grams will be monitored while lying on a pressure sensitive mat.
  Interventions: Device: Pressure sensitive mat
- Incubator + 1500 - 2500 g: Infants currently in an incubator with a weight between 1500 - 2500 grams will be monitored while lying on a pressure sensitive mat.
  Interventions: Device: Pressure sensitive mat
- Overhead warmer + <1500 g: Infants currently in an overhead warmer with a weight less than 1500 grams will be monitored while lying on a pressure sensitive mat.
  Interventions: Device: Pressure sensitive mat
- Overhead warmer + 1500 - 2500 g: Infants currently in an overhead warmer with a weight between 1500 - 2500 grams will be monitored while lying on a pressure sensitive mat.
  Interventions: Device: Pressure sensitive mat
- Overhead warmer + >2500 g: Infants currently in an overhead warmer with a weight over 2500 grams will be monitored while lying on a pressure sensitive mat.
  Interventions: Device: Pressure sensitive mat
- Crib + 1500 - 2500 g: Infants currently in a crib with a weight between 1500 - 2500 grams will be monitored while lying on a pressure sensitive mat.
  Interventions: Device: Pressure sensitive mat
- Crib + >2500 g: Infants currently in a crib with a weight over 2500 grams will be monitored while lying on a pressure sensitive mat.
  Interventions: Device: Pressure sensitive mat

INTERVENTIONS:
Device: Pressure sensitive mat — Infant placed on pressure sensitive mat and has physiological parameters recorded.

SUMMARY:
This is a pilot study that provides the investigators with an opportunity to assess the application of PSM technology for patient monitoring in the NICU. This is a prospective, observational, cohort study.The investigators expect the duration of infant participation in this study to be 6 hours per single recording session with no follow-up required.

DETAILED DESCRIPTION:
Study Procedures/Evaluations

* The trial will be conducted at the CHEO NICU. The non-invasive patient monitoring equipment that has no direct contact with infant's skin, includes a pressure sensitive mat (PSM) from the LX100 series (XSensor Technology Corp. Calgary, Canada, XSensor.com) and a video camera.
* The patient will be lying in an incubator, on an overhead warmer neonatal bed, or an open crib (whatever bed type they are currently being nursed in/on). The patient's nurse will place the PSM on the mattress and under the patient's bedsheet where it will have no contact whatsoever with the patient. The PSM placement under the infant will happen at a time when the infant would normally be handled/moved.
* Data from the following four sources will be recorded simultaneously in each session:

  1. Contact pressure data from PSM
  2. Physiologic monitor data including blood oxygen saturation (SpO2), heart rate (HR), pulse rate (PR), respiratory rate (RR), and the alarms associated with each of these physiologic data streams. This data is collected from monitors that the patient has attached as part of their usual care.
  3. Video of the patient
  4. Event annotations collected by a bedside research assistant on a PC, laptop or tablet.
* All data will be de-identified using unique study identifiers. The NICU research team will assign these study identifiers and keep this information on a Master Study List separate from all recorded data.
* The PSM connects to an X3 Pro Sensor Pack that feeds into an X3 Pro Electronic Platform that is connected via USB to a laptop running the X3 Pro software. The X3 Pro software is used to record PSM data and video simultaneously. The PSM is powered from an approved AC power supply and is connected to the data acquisition computer via USB. The XSensor PSM system is already being used with adult patients, however, the electrical safety of our final configuration will also be established through independent inspection (see below). The pressure mat will be covered by one or more bedsheets at all times. The baby will not be permitted to come in contact with the mat to reduce the risk of electrical shock and airway obstruction.
* Bench tests will be conducted by CHEO Clinical Engineering to confirm that leakage current measurements from the mat and the entire system will meet the limits published in Requirement EN60601. If any deficiencies are identified alternations to the system will then be completed prior to a special inspection by Canadian Standards Association (CSA). A special electro medical inspection will be arranged with CSA for the final configuration of PSM, laptop, and power supplies.
* The video camera will be mounted on a tripod to capture patient movements, routine care, and clinical interventions if any. We will capture the entire body, the head being very important as this is where most interventions occur such as nasal gavage feeding, ventilator support and airway suctioning. Video analysis has shown to be particularly useful for estimating RR in neonates [39].
* A bedside research assistant (RA) will manage all data recordings on a computer kept by the patient's bedside for up to 6 hours per recording session.
* Physiologic data including the patient's heart rate (HR), respiratory rate (RR), oxygen saturation levels (SpO2) and pulse rate (PR) as well as corresponding alarms for each data stream shall be logged from the bedside Dräger patient monitor onto a computer.
* The RA will simultaneously annotate all patient events including movements, routine care, and clinical interventions on an electronic device such as a PC, laptop, or tablet.
* The RN who will respond to the alarms will be asked for their clinical opinion as to the veracity (artifact or clinically important) of the alarms and this opinion will be annotated by the RA.

ELIGIBILITY:
Inclusion Criteria:

* Infants in the NICU will be eligible if their parents speak English or French and can be approached for consent.

Exclusion Criteria:

* Patients who are moribund, suspected of having a neuromuscular condition affecting their movement or who are receiving muscle relaxant medications will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants in the NICU will be eligible if their parents speak English or French and can be approached for consent.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of information collected from pressure sensitive mat. | Six hours
  This study will examine the potential for incorporating PSM and video data analysis as part of an integrated patient monitoring environment.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Harrold, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No